CLINICAL TRIAL: NCT04072809
Title: Dissecting the Genetics of Fetal Alcohol Spectrum Disorders
Acronym: DiGFASD
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tatiana Foroud, Joe C. Christian Professor of Medical & Molecular Genetics, Indiana University
Other Study IDs: 1801900355; U01AA026103 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: Fetal Alcohol Syndrome; Alcohol Related Neurodevelopmental Disorder; Alcohol-Related Birth Defects; FAE (Fetal Alcohol Effects); FASD; Partial Fetal Alcohol Syndrome; ND-PAE; Prenatal Alcohol Exposure; fetal exposure to ethanol during pregnancy; FAS
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All participants in the study will experience the same procedures.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study does not involve any interventions.

SUMMARY:
The purpose of this study is to help scientists understand why some people who were exposed to alcohol in the womb have special facial features but other people do not. This study will test if genetics (or DNA) explains these differences. We hope this will help improve treatments and interventions for people with fetal alcohol spectrum disorders (FASD).

Participants in this study (or their parents or legal guardians) will be asked to:

* Answer some questions about themselves. These questions ask about their demographic background (such as gender, race, ethnicity, income, and education), their health history, and their mother's health during her pregnancy with them (if that information is known).
* Speak with study staff briefly by phone or video chat to confirm enrollment in the study and ask any questions they have.
* Take photographs of their face.
* Provide a saliva sample for genetic research.

Participants can complete the study at home from anywhere in the world. The questions can be answered online, over the phone, or on paper. Adopted families are welcome to enroll. The study pays for all shipping costs.

DETAILED DESCRIPTION:
Fetal Alcohol Syndrome (FAS) typically involves poor growth for age, particular facial characteristics, and cognitive deficiencies. Although FAS was first described in the literature over 40 years ago, significant challenges remain in the development of rapid and efficient approaches to identify individuals who were prenatally exposed to alcohol. Further, no widely available effective interventions or treatments to improve the long term outcomes of individuals with FAS and related disorders (collectively known as Fetal Alcohol Spectrum Disorders or FASD) exist, despite the high prevalence (as high as 33.5 per 1,000 in some communities) of FASD across the United States.

The Collaborative Initiative on Fetal Alcohol Spectrum Disorders (CIFASD) seeks to address critical issues related to earlier and improved recognition of FASD, identify biomarkers of exposure, and elucidate the genetic risk factors contributing to FASD risk and resilience by conducting multidisciplinary projects and maintaining cooperative resources. This project is part of CIFASD's ongoing efforts and will specifically address the elucidation of genetic factors that contribute to risk and resilience in FASD.

Prior work with animal models of FASD have identified genetic variants that contribute to alterations in facial morphology after exposure to alcohol during embryonic development (McCarthy et al., 2013). Prenatal alcohol exposure also activates immune pathway genes in animal models. The identification of these genetic factors suggest that genetic variation may similarly contribute to differences in response to prenatal alcohol exposure in humans. The goal of this project is to identify genetic variants that protect against or increase the effects of prenatal alcohol exposure in humans.

ELIGIBILITY:
Inclusion Criteria:

* Documented or suspected history of prenatal alcohol exposure OR Fetal Alcohol Spectrum Disorder (FASD) diagnosis
* Speaks English

Exclusion Criteria:

* No documented or suspected history of prenatal alcohol exposure OR FASD diagnosis
* Does not speak English

Ages: 1 Month to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with FASD or prenatal alcohol exposure will be recruited throughout the world.
Sampling Method: Non-Probability Sample
Enrollment: 751 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Facial Risk Score | through study completion, an average of 1 year
  Facial Risk Score
  Each participant's facial images will be evaluated and a Facial Risk Score will be assigned to each individual. This risk score is relative to all individuals participating in the study, and therefore will be updated at the end of each year. Final scores will be completed at the end of the study. The risk score is computer-based, with high scores indicating increased dysmorphology and low scores indicating decreased dysmorphology.
Whole Exome Sequencing (WES) | through study completion, an average of 1 year
  Whole Exome Sequencing
  After Facial Risk Scores have been assigned to each individual, two subsets of the study population will be selected: those with high risk scores, and those with low risk scores. Saliva samples from these subpopulations will be subjected to Whole Exome Sequencing (WES). Rare variant analysis will be performed in each gene to evaluate whether there are more rare variants in individuals from one group (e.g., high risk scores) compared to the other group (e.g., low risk scores). This will enable us to determine if the variant increases risk (more common in those with high risk scores) or increases resilience (more common in those with low risk scores).

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Foroud, Principal Investigator — Indiana University; Leah Wetherill, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The types of information that will be shared include facial images and derived data, genetic data, demographic data, and data related to FASD diagnoses or prenatal alcohol exposure. No personally identifying information (such as name or birthdate) other than facial images will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: indefinite
Access Criteria: Researchers who would like to access IPD must apply for access through the Collaborative Initiative for Fetal Alcohol Spectrum Disorders (CIFASD).
URL: https://cifasd.org

REFERENCES:
- See also: The DiGFASD study web portal for enrolling in and learning about the study. — https://digfasd.org